CLINICAL TRIAL: NCT01174056
Title: Noninvasive Quantification of the Pulmonary Anti-inflammatory Effect of Rosiglitazone
Brief Title: Evaluation of Rosiglitazone Anti-inflammatory Effect With FDG-PET Imaging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DDCF-2010060
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Lung Inflammation
Keywords: Lung inflammation; positron emission tomography; fluorodeoxyglucose; rosiglitazone; zileuton; lung anti-inflammatory therapy
MeSH Terms: conditions — Pneumonia | interventions — zileuton; Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pioglitazone+zileuton placebo (Experimental): Pioglitazone 45 mg qD for 2 weeks plus Sugar pill q6hr for 5 days
  Interventions: Drug: Zileuton placebo; Drug: Pioglitazone
- Zileuton+pioglitazone placebo (Experimental): Sugar pill qD for 2 weeks plus Zileuton 600 mg q6hr for 5 days
  Interventions: Drug: Zileuton; Drug: Pioglitazone placebo
- Pioglitazone placebo+zileuton placebo (Sham Comparator): Sugar pill qD for 2 weeks plus Sugar pill q6hr for 5 days
  Interventions: Drug: Pioglitazone placebo; Drug: Zileuton placebo

INTERVENTIONS:
Drug: Zileuton — 600 mg tablets po QID for 5 days prior to endotoxin, stopping 24 hours after endotoxin instillation
  Other Names: Zyflo
  Arms: Zileuton+pioglitazone placebo
Drug: Pioglitazone placebo — Lactose filled gelatin capsule, size 00, 1 tablet po bid x 2 weeks prior to endotoxin instillation until 24 hours after endotoxin.
  Arms: Pioglitazone placebo+zileuton placebo; Zileuton+pioglitazone placebo
Drug: Zileuton placebo — Placebo tablets provided by manufacturer of Zyflo CR (Cornerstone Therapeutics), 2 tablets po bid x 5 days prior to endotoxin instillation until 24 hours after endotoxin.
  Arms: Pioglitazone placebo+zileuton placebo; Pioglitazone+zileuton placebo
Drug: Pioglitazone — PPAR-gamma agonist
  Other Names: Actos
  Arms: Pioglitazone+zileuton placebo

SUMMARY:
The purpose of this research study is to gain understanding of the basic responses of the lung to inflammation and specifically if a certain medication can reduce the inflammation alone or in combination with another. Inflammation is the way our bodies react to irritation or injury, and involves red, warm, and often painful swelling of the affected tissue. "Acute lung injury" involves inflammation that is not specific to one area of the lung and is caused by any one of several conditions: infection, trauma, breathing toxic substances, etc. When lung injury is severe, not enough oxygen can get into the body; this can lead to the need for mechanical support of breathing (mechanical ventilation), problems with brain, heart or other organ function, and in some cases, death.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman, any race or ethnicity, age 19 - 44 years old
* Screening FEV1 and FVC > 90% of predicted
* Screening oxygen saturation by pulse oximetry >97% on room air
* Capable of lying still and supine within the PET/CT scanner for ~1.5 hours
* Capable of following instructions for breathing protocol during CT portion of PET/CT
* Able and willing to give informed consent
* BMI < 35

Exclusion Criteria:

* Pregnancy (confirmed by qualitative urine hCG pregnancy test)
* Lactation
* Active menstruation
* History of cardiopulmonary disease
* Currently taking any prescription medications
* History of tobacco use or illicit drug use within the past year
* Presence of implanted electronic medical device
* Enrollment in another research study of an investigational drug
* Known allergy to rosiglitazone or zileuton
* Known allergy to both trimethoprim/sulfamethoxazole and amoxicillin
* Known allergy to drugs routinely used during bronchoscopy
* History of chronic active liver disease or acute liver disease within the past 3 months
* SGOT >47 IU/L, SGPT > 53 IU/L, or bilirubin > 1.1 mg/dl
* Inability lie flat for 1.5 hours for PET/CT scans or follow breathing protocol instructions for the CT portion of the PET/CT
* Prior research-related radiation exposure within the past year such that participation in this study would result in exposures that exceed the limits as defined by the FDA RDRC regulations (21 CFR 361.1).

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Ki, measure of FDG uptake | Before and after endotoxin
  Ki will be measured before and after endotoxin. Primary outcome measure is change in Ki (post- minus pre-endotoxin value) and absolute Ki after endotoxin.

SECONDARY OUTCOMES:
Bronchoalveolar lavage (BAL) fluid cell counts | After endotoxin
  Total and neutrophil cell counts obtained by bronchoalveolar lavage after endotoxin.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine L Chen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University / Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Chen DL, Huang HJ, Byers DE, Shifren A, Belikoff B, Engle JT, Arentson E, Kemp D, Phillips S, Scherrer DE, Fujiwara H, Spayd KJ, Brooks FJ, Pierce RA, Castro M, Isakow W. The peroxisome proliferator-activated receptor agonist pioglitazone and 5-lipoxygenase inhibitor zileuton have no effect on lung inflammation in healthy volunteers by positron emission tomography in a single-blind placebo-controlled cohort study. PLoS One. 2018 Feb 7;13(2):e0191783. doi: 10.1371/journal.pone.0191783. eCollection 2018. PMID 29414995